CLINICAL TRIAL: NCT06715618
Title: The Use of the Functional Movement Screen™ in Preventing Injuries in Amateur Rugby Players: a Longitudinal Prospective Study
Brief Title: The Use of the Functional Movement Screen™ in Preventing Injuries in Amateur Rugby Players
Acronym: FMSrugbyAMA
Status: Recruiting | Type: Observational
Sponsor: Hopital La Musse (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A01804-43
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Prevention; Risk; Injuries; Rugby; Rugby Player
Keywords: Amateur Rugby; Prevention; Risk; Injuries; Players
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FMS group: Each participant will perform two FMS™, one at the beginning of the competitive season and one at the end of the competitive season. The test will take 30 minutes per player. The initial interview will last 20 minutes. Players will also be monitored throughout the season to collect all injuries sustained by the participants in the study.
  Interventions: Other: FMS test

INTERVENTIONS:
Other: FMS test — Each participant will perform two FMS™, one at the beginning of the competitive season and one at the end of the competitive season. The test will take 30 minutes per player. The initial interview will last 20 minutes. Players will also be monitored throughout the season to collect all injuries sustained by the participants in the study.

SUMMARY:
Rugby is a team contact sport that demands unparalleled physical engagement. This practice, which combines random running patterns with changes in speed and direction, also involves frequent contact situations with other players. These phases of the game account for 48% to 80% of total injuries. Injury prevention is an integral part of the physical therapist's expertise and plays a crucial role in reducing the occurrence of musculoskeletal injuries and mitigating their devastating consequences.

The implementation of a risk prevention tool is particularly relevant for a population prone to injuries. However, the practicality of such a tool must be considered, as adherence to an injury prevention program depends on the "perceived usefulness, intensity, and time investment of the program".

One tool appears to meet these criteria: the Functional Movement Screen™ (FMS™). This tool is designed to "evaluate an individual's functional movement patterns" and, according to its authors, can serve as "a crucial tool" for returning to sports after an injury or a period of inactivity. Given the high incidence of injuries in rugby players, calculating the injury incidence in this population and correlating it with FMS™ scores could provide valuable insights.

For this prospective study, forty amateur rugby players from various clubs in Normandy competing at the Federal 3 level will be recruited using a recruitment letter and a call for volunteers.

Each participant will perform two FMS™ (7 movements), at the beginning of the competitive season and at the end of the competitive season. The test will last 30 minutes per player. The initial interview will last 20 minutes. There will also be a follow-up of the players throughout the season to collect all injuries sustained by participants in the intervention.

The main expected outcome is a significant correlation (p < 0.05) between the FMS™ score and injury incidence. This correlation may then indicate a good predictive capacity of the FMS™, allowing it to be considered a predictive tool for injury risk.

To evaluate the correlation between two variables (injury incidence sustained by the player and the FMS™ score), the Spearman correlation coefficient will be used. This coefficient, if its value approaches -1 or 1, will indicate a good correlation between the player's injury incidence and their FMS™ score. Conversely, if the coefficient approaches 0, the correlation will be considered poor.

In a second phase, it is expected that a competitive season will directly affect the FMS™ score, highlighting the difficulty for an amateur player to maintain their physical capacities throughout an entire season.

ELIGIBILITY:
Inclusion Criteria:

* Players licensed with the French Rugby Federation (FFR): Their affiliation with the FFR requires a medical certificate confirming no contraindication to competitive sports practice.
* Players aged at least 18 years old, legally adults.
* Healthy players who have not sustained any musculoskeletal injuries or undergone surgical interventions in the past 6 months.
* Players competing in "Fédérale 3."
* Players from clubs based in Normandy.

Exclusion Criteria:

* Minor players
* Female players
* Players injured during the first interview or the first FMS™
* Players who are or have been professional athletes
* Players with a history of frequent serious injuries that could pose a risk to their continued participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The chosen study population consists of amateur rugby players from Normandy. Forty rugby players will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-05-03 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The FMS™ score | At the beginning and the end of the enrollment (8month after enrollment)
  The Functional Movement Screen™ (FMS™) is a tool designed to "evaluate an individual's functional movement patterns" and, according to its authors, can represent "a crucial tool" for returning to sport after an injury or a break from sports. It consists of an assessment of seven so-called fundamental movements, which require good neuromuscular and motor control, as well as balance and stability. These movements aim to place the evaluated subject in extreme positions to highlight significant imbalances throughout the body. This test consists of a score from 0 to 3 for each of the 7 movements, and a final score out of 21 points. The FMS reveals functional deficits by highlighting compensatory movements. The higher the score, the fewer compensatory movements.

SECONDARY OUTCOMES:
The number of injuries | From enrollment to the end of study (8months)
  The secondary endpoint is the number of injuries. An injury is defined as "any physical complaint caused by an energy transfer exceeding the body's ability to maintain its structural and/or functional integrity, sustained by a player, regardless of the need for medical treatment or the time lost due to the injury". Here, only injuries involving time lost, the "time-loss injury," are considered. Therefore, in this study, a player is considered injured if they are unable to participate in the following training session or match due to the injury. Any other inability, such as personal or professional reasons, will not be considered. This method of data collection is widely used in sports medicine due to its simplicity, even when athletes themselves report the injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: Undecided